CLINICAL TRIAL: NCT00195585
Title: Post-Approved Phase III Study of 1-LV/5FU Therapy
Brief Title: Study Evaluating Isovorin in Colon Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ISO/5FU-11
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2009-08-13 (Estimated); Status verified 2009-08

CONDITIONS: Colon Cancer
Keywords: Colon Cancer
MeSH Terms: conditions — Colonic Neoplasms | interventions — Leucovorin

INTERVENTIONS:
Drug: Isovorin
Drug: UFT

SUMMARY:
The purpose of the study is to verify superiority of 1-LV/5FU therapy to UFT Therapy of relapse-free survival time in patients with Dukes C and Cure A colon cancer. Secondary endpoints include disease-free survival time, survival time, and safety.

ELIGIBILITY:
Inclusion Criteria:

* Dukes C, Cure A colon cancer diagnosed histologically or cytologically
* Normal organ function of bone marrow, heart, liver and kidney
* Age 20-75

Other inclusion applies

Exclusion Criteria:

* Serious bone marrow suppression, infection, heart disease or complication
* Familial adenomatous polyposis or hereditary nonpolyposis
* Pregnant or breastfeeding women

Other exclusion applies

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 650
Dates: Start 2002-10; Primary Completion 2006-02 (Actual); Study Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
Relapse-free survival time

SECONDARY OUTCOMES:
Disease-free survival time, survival time, safety

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (1):
- Tokyo, Japan